CLINICAL TRIAL: NCT04143282
Title: Evaluation of the Effect of Metformin on Metastatic Breast Cancer as Adjuvant Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hager salah el din (Other)
Responsible Party: Sponsor-Investigator, Hager salah el din, pharmacist, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWA00015574/6-01-2019/korany
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Breast Cancer
Keywords: metformin; non metastatic breast cancer; non-diabetic
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin group (Experimental): Non Diabetic metastatic breast cancer Patients will take metformin 1 gm. twice daily (Nathan 2009) along with standard chemotherapy
  Interventions: Drug: Metformin plus chemotherapy
- control group (Other): Non Diabetic metastatic breast cancer Patients will take standard chemotherapy only
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Metformin plus chemotherapy — determine the effect of metformin along with standard chemotherapy
  Arms: Metformin group
Drug: Chemotherapy — standard chemotherapy
  Arms: control group

SUMMARY:
This study aims to determine the effect of metformin along with standard cancer treatment, and its effect on the prognosis of the metastatic breast in non-diabetic patients.

DETAILED DESCRIPTION:
the role of metformin when combined with traditional metastatic breast cancer treatment in non-diabetic patients compared to diabetic patients who are not using metformin. In this randomized control study, there will be a demonstration either it is effective to suppress tumor burden or not through normal screening for tumor.

ELIGIBILITY:
Inclusion Criteria:

* The non-diabetic patients will be included in the study if they meet the following criteria:

  1. Confirmed metastatic breast cancer (IV stage) radiologically or by clinical evaluation receiving chemotherapy
  2. Age between 18- 70 years.
  3. Life expectancy at least 6 months

Exclusion Criteria:

* The patients will be excluded from the study if they have the following criteria:

  1. Bad prognosis disease: Criteria defined as the following

     * If patient >70 years
     * If patient has bad site metastasis (brain)
  2. Hypersensitivity for metformin: if happened patient will be treated as following

     • Pheniramine Maleate 3 times daily for 7 days and Tablet Dexamethasone 1mg daily in 2 divided doses for 5 days [16].
  3. Any condition associated with increased risk of metformin-associated lactic acidosis (e.g., congestive heart failure defined as New York Heart Association {NYHA} Class III or IV functional status; the history of acidosis of any type, severe infections, kidney or liver disease, respiratory disease, seizures .
  4. Diabetic patients.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — metastatic breast cancer female
Enrollment: 250 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
The radiologic response rate | 3 months
  The Response Evaluation Criteria in Solid Tumors (RECIST 1.1) was used to evaluate the response to chemotherapy alone in case of control arm and chemotherapy plus metformin in case of drug arm for breast cancer with distant metastasis
Overall survival (OS) | 6 months
  the time period from the start of trial till death or end of follow-up
Progression-free survival | 6 months
  from the time between start of the trial and recurrence or disease progression, or end of follow-up

SECONDARY OUTCOMES:
Insulin Growth like Factor -1 (IGF-1) at base line and after 3 cycle. | 3 months
  measure blood Insulin Growth like Factor -1 (IGF-1) at the begining of trial then after 3 months at the end of 3 cycles (each cycle arround 28 days )

CONTACTS AND LOCATIONS:
Overall Officials: ahmed a berry, PhD, Study Director — Faculty of Medicine, Beni Suef University; ahmed h shaaban, MD, Study Director — Faculty of Medicine, Beni Suef University; hoda m rabea, PhD, Study Director — Faculty of pharmacy, Beni Suef University
Locations (1):
- Beni-Seuf University Hospital, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Yes
upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 MONTHS
Access Criteria: hager.salah@rocketmail.com

REFERENCES:
- [Derived] Salah H, Rabea H, Sheemy MS, Rabie AI, Moustafa HAM, Elberry AA, Hassan A. Targeting insulin-like growth factor-1 (IGF-1) by using metformin in non-diabetic metastatic breast cancer female patients: a randomized controlled trial. Cancer Chemother Pharmacol. 2025 Jun 28;95(1):64. doi: 10.1007/s00280-025-04791-8. PMID 40579605